CLINICAL TRIAL: NCT00886223
Title: Laparoscopic Sacropexy: Clinical Prospective Study With Robot-Assisted Technique(da Vinci®-System)
Brief Title: Laparoscopic Sacropexy With Robot-Assisted Surgical System
Acronym: RobPex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Dimitri Sarlos,M.D, Vice chairman, Department of Gynecology and Obsterics, Kantonsspital Aarau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSA-RobPex1
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Vaginal Vault Prolapse
Keywords: vaginal vault prolapse repair; robot-assisted laparoscopic sacropexy; robot-assisted laparoscopic sacrocolpopexy; robotic laparoscopic sacropexy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: laparoscopic robot-assisted sacropexy

INTERVENTIONS:
Procedure: laparoscopic robot-assisted sacropexy — Repair of vaginal vault prolapse with laparoscopic sacropexy assisted by robotic surgical system (da Vinci®-System)
  Other Names: robotic laparoscopic sacropexy; robot-assisted laparoscopic sacrocolpopexy; robotic laparoscopic sacrocolpopexy

SUMMARY:
The aim of the study is to evaluate safety and outcome of robot-assisted laparoscopic sacropexy regarding perioperative data, objective anatomical results and postoperative quality of life.

DETAILED DESCRIPTION:
Vaginal vault prolapse is a common finding in Gynecology. Many different approaches for vaginal vault prolapse repair are available. During the last few years robot-assisted surgery has been introduced in many surgical specialties and experiences in gynecologic surgery are very limited.

Several aspects like the wider range of motion of robot-instruments leading to more precision in surgery, the 3 dimensional optical system and the ergonomically designed console may offer some advantages. For better judgment these possible benefits as well as safety and outcome need to be evaluated and compared with conventional laparoscopic sacropexy techniques.

This prospective clinical study evaluates robot-assisted laparoscopic sacropexy (da Vinci®-System) focusing on peri-operative data, objective anatomical results and postoperative quality of life and compares the results with conventional laparoscopic sacropexy. Pre- peri- and post-operative data are collected using the prolapse quantification system (POP-Q) and the German Pelvic Floor questionnaire. The objective of the study will be to investigate if the robot assisted procedure shows significant advantages for the patient considering duration of surgery, complications, hospitalization, quality of life and costs.

ELIGIBILITY:
Inclusion Criteria:

* vaginal vault prolapse
* recurrence after vaginal prolapse repair
* signed consent

Exclusion Criteria:

* rectocele
* BMI > 40

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery | during hospitalisation

SECONDARY OUTCOMES:
Complications | 6 months after hospitalisation
Anatomical results | 6 months after hospitalisation
Quality of life | 6 months after hospitalisation
Costs | 6 months after hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Sarlos, MD, Study Chair — Kantonsspital Aarau, Department of Obsterics and Gynecology
Locations (1):
- Kantonsspital Aarau, Aarau, Switzerland